CLINICAL TRIAL: NCT06768736
Title: Randomised Controlled Trial on an Early Warning System for Allergic Rhinitis in the MASK-air® App
Brief Title: Early Warning System for Allergic Rhinitis in the MASK-air® App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Universidade do Porto; 101057131 (Other Grant/Funding Number: Horizon Europe research and innovation framework programme)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Generic messages already delivered by MASK-air® (No Intervention)
- Early warning system personalised forecasting messages (Experimental)
  Interventions: Combination Product: Personalised early warning system

INTERVENTIONS:
Combination Product: Personalised early warning system — Early warning system personalised forecasting messages
  Arms: Early warning system personalised forecasting messages

SUMMARY:
The primary objective consists in the comparison of the combined symptom medication score values between (i) patients randomised to the early warning system personalised forecasting messages, and (ii) patients randomised to generic messages already delivered by MASK-air®.

The combined symptom medication score has recently been developed in a data-driven way and validated (https://eaaci.org/images/CSMS.pdf); it assesses allergic rhinitis control taking into account both reported symptoms and medication use.

As secondary objectives, visual analogue scales on allergic rhinitis symptoms (VAS global, nasal, eye, asthma), and medication use will also be separately compared.

DETAILED DESCRIPTION:
In patients with allergic rhinitis, forecasting potential exacerbation of symptoms may allow patients to adopt the most adequate preventive measures. In this context, we are developing an early warning system combining atmospheric, pollen, patient symptoms and online activity data.

This early warning system will be incorporated in a mobile health app, and aims to provide patients with messages indicating whether exacerbations are expected in the subsequent five days.

To test the effectiveness of the early warning system in avoiding a worsening of patients' symptoms, undertaking a randomised controlled trial is warranted, particularly comparing personalised forecasting messages versus generic messages.

The clinical study will assess an early warning system, which will be developed through the CATALYSE project. This early warning system will be incorporated in MASK-air®, a mobile health app implemented in 19 European countries, and which allows for patients to register their daily allergic rhinitis symptoms(rhinitis, conjunctivitis and asthma) and medication. The early warning system will be based on: patients' symptom information (as registered in MASK-air®); and atmospheric and pollen forecasts provided by SILAM model and Copernicus systems (which are able to provide forecasts for six main allergic pollen types in Europe, and is able to assimilate new observations registered with an hourly time resolution).

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (≥18 years old) of both sexes with clinical diagnosis of allergic rhinitis according to ARIA associated with pollen allergy.

Exclusion Criteria:

* Illiterate patients
* Patients without smartphone
* Patients who are not able to complete a daily monitoring questionnaire on allergic rhinitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Combined symptom medication score values | From enrollment to the end of intervention at 2 weeks
  Daily symptom and medication data provided by patients allow the calculation of two validated daily combined symptom-medication scores from formulae previously published:
  * the CSMS (combined symptom-medication score)
  * e-DASTHMA.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided